CLINICAL TRIAL: NCT06025162
Title: Evaluation of Chemical Venous Thromboembolism Prophylaxis in Trauma
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 028.PHA.2022.D
Record Dates: First submitted 2022-12-20; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Thromboembolism, Venous
MeSH Terms: conditions — Venous Thromboembolism | interventions — Enoxaparin; Contraindications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LMWH dosing strategies: MDMC's trauma VTE prophylaxis guideline will be used to classify patients into two treatment arms ("weight-based" or "standard dose") based on their dose of enoxaparin at 48 hours post-VTE prophylaxis initiation
  Interventions: Drug: enoxaparin

INTERVENTIONS:
Drug: enoxaparin — dose of enoxaparin at 48 hours post-VTE prophylaxis initiation
  Other Names: Accessing for contraindication for chemical VTE prophylaxis

SUMMARY:
Venous thromboembolism (VTE) causes up to 100,000 deaths annually. Between 10%-30% of patients die within one month of VTE diagnosis, while survivors remain at increased risk for VTE recurrence or other complications like post-thrombotic syndrome or chronic pulmonary hypertension in the following decade. Trauma patients have many risk factors that predispose them to a VTE. During the first 48 hours after blunt trauma, patients are prothrombotic due to the release of procoagulant factors, have excessive thrombin generation due to extensive tissue and vascular injury, and have reduced circulation of endogenous anticoagulants like protein C.

DETAILED DESCRIPTION:
Trauma patients have many risk factors that predispose them to a VTE. During the first 48 hours after blunt trauma, patients are prothrombotic due to the release of procoagulant factors, have excessive thrombin generation due to extensive tissue and vascular injury, and have reduced circulation of endogenous anticoagulants like protein C. Trauma patients are immobile for prolonged periods of time due to frequent surgical intervention and extended sedation. Even when administered chemoprophylaxis, up to 15% of trauma patients develop thromboses. Given the high rates of thromboses, one study validated certain risk factors for VTE among trauma patients. This study categorized patients as high-risk or very high-risk of VTE based on patient-specific factors. High-risk factors for VTE included a history of VTE, repair or ligation of major venous injury, an abbreviated injury scale (AIS) >2 for the head, a Glasgow coma Scale (GCS) score <8 for >4 hours after trauma, and age ≥60 years. Very high-risk factors for VTE consist of complex lower extremity fractures, pelvic fractures, spinal cord injury with associated para- or quadriplegia, and age ≥75 years. The 2020 Western Trauma Association guidelines recommend initiation of VTE prophylaxis with enoxaparin within 24 hours of admission in trauma patients, with special consideration for patients with active bleeding, solid organ injury, traumatic brain injury (TBI), or spinal cord injury. Several studies support this recommendation and correlate delays in VTE prophylaxis initiation and interruption in therapy with increased risk of VTE.

Recent evidence also highlights that the standard trauma VTE dosing strategy of 30 mg of enoxaparin twice daily often fails to reach adequate target anti-Xa levels in trauma patients. Thus, consideration of 0.5 mg/kg enoxaparin twice daily with adjustments based on anti-Xa levels may be considered in patients at highest risk of VTE. This strategy may be associated with improved outcomes while mitigating adverse effects like clinically significant bleeding.

Despite these recommendations, providers may choose to delay initiation of VTE prophylaxis due to a patient's apparent bleeding risk. Trauma-induced coagulopathy is present in 20%-25% of patients and is associated with a higher incidence of bleeding, increased transfusion requirements, and elevated risk of multi-organ failure versus patients without this coagulopathy. Additionally, chemical VTE prophylaxis with anticoagulants like LMWH may increase bleeding possibility, especially in patients that are at risk for emergent surgical intervention. Even so, current evidence supports that early initiation of VTE prophylaxis in high-risk patients, as benefit outweighs bleed risk.

Special trauma populations like TBI, spinal cord injury, and solid organ injury have been the focus of recent studies evaluating bleeding risk after initiation of VTE prophylaxis. In one study, TBI patients were at a significantly increased risk for VTE and substantial delays in VTE prophylaxis initiation (7 days vs 1.5 days) versus non-TBI patients. Concern for intracranial hemorrhage (ICH) progression was most likely found to cause delays in VTE prophylaxis in this high-risk population despite the overall low incidence of this finding.15 In patients with intracranial bleeding, two studies identified that initiation of VTE prophylaxis 24 hours after stable computerized tomography (CT) imaging did not increase risk of ICH progression while decreasing overall incidence of VTE. For patients with blunt solid organ injury, initiation of VTE prophylaxis within 48 hours of injury was not associated with an escalation in bleeding events, but delaying prophylaxis beyond 72 hours correlated with in increased risk for VTE. VTE prophylaxis initiation within 48 hours of non-operative spinal cord injury was also found to significantly reduce VTE incidence versus initiation beyond 48 hours.

In 2020, Methodist Dallas Medical Center's (MDMC's) pharmacy department developed a guideline for VTE prophylaxis in trauma patients. This document was designed to improve patient outcomes by providing evidence to assist providers when initiating patients on chemical VTE prophylaxis and support the safe and efficacious use of weight-based VTE prophylaxis regimens in patients at high-risk of VTE. The guideline's algorithm first recommends assessing for contraindications for chemical VTE prophylaxis (like ongoing hemorrhagic shock). After assessing contraindications and creatinine clearance, the document provided guidance on LMWH dosing strategies, suggested patient populations for weight-based prophylaxis regimens, and recommended timeframes for initiation of VTE prophylaxis based on injury type. Patient outcomes have not been assessed since the implementation of MDMC-specific VTE prophylaxis trauma guidelines.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Admitted to the trauma service between October 1,2021 and March 31, 2022
* Weight ≥50 kg
* Received chemical VTE prophylaxis with LMWH for at least 48 hours
* At "high risk" or "very high risk" of VTE8

Exclusion Criteria:

* Death, discharge, or hospice within 48 hours of admission
* Documented heparin allergy (heparin-induced thrombocytopenia)
* Indication for therapeutic anticoagulation, either prior to admission or during hospitalization
* Prisoners
* <18 years of age
* Pregnancy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective observational cohort study involving patients admitted to the trauma service at Methodist Dallas Medical Center between October 1, 2021 and March 31, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Episodes of clinically significant bleeding after VTE prophylaxis initiation | "48 Hours"
  High-risk factors for VTE included a history of VTE, repair or ligation of major venous injury, an abbreviated injury scale (AIS) >2 for the head, a Glasgow coma Scale (GCS) score <8 for >4 hours after trauma, and age ≥60 years. Very high-risk factors for VTE consist of complex lower extremity fractures, pelvic fractures, spinal cord injury with associated para- or quadriplegia, and age ≥75 years.
Time to clinically significant bleeding after VTE prophylaxis initiation | "48 Hours"
  During the first 48 hours after blunt trauma, patients are prothrombotic due to the release of procoagulant factors, have excessive thrombin generation due to extensive tissue and vascular injury, and have reduced circulation of endogenous anticoagulants like protein C.5,6 Trauma patients are immobile for prolonged periods of time due to frequent surgical intervention and extended sedation.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Reiter, PharmD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center Pharmacy, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No